Effects of transcutaneous electrical nerve stimulation for the treatment of pain and respiratory function following mastopexy with augmentation. Study protocol for a randomized controlled trial

## Statistical methods for primary and secondary outcomes.

- The Kolmogorov–Smirnov (KS) normality test will be applied to evaluate the distribution of data obtained for the variables (pain intensity at rest, pain intensity during movement, pain intensity during maximum inspiratory pressure, pain intensity during maximum expiratory pressure and vital capacity) at the four assessments (T0, T1, T2 and T3). Data with normal distribution will be expressed as mean and standard deviation and those with non-normal distribution will be expressed as median and interquartile range. Either ANOVA or the Kruskal-Wallis test will be used for the inter-group and intra-group comparisons of the variables of interest, depending on the distribution of the variables.
- Repeated-measures two-way ANOVA and the Holm-Sidak post hoc test will be used for comparisons among evaluation times for quantitative variables with a normal homogeneous distribution.
- The significance level will be set at p<0.05 for all statistical tests. The data will be analyzed using the SPSS software (v.17; SPSS Inc; Chicago, IL, USA) by an investigator blinded to the allocation of the participants to the different groups.